CLINICAL TRIAL: NCT07095972
Title: Optimizing Glycemic Control in Metabolic Surgery With Continuous Glucose Monitoring
Brief Title: Continuous Glucose Monitoring in Metabolic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: LA CaTS Clinical Research Resources Core (Unknown)
Responsible Party: Principal Investigator, Yun Shen, Assistant professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-021-PBRC
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Obesity (Disorder)
Keywords: Diabetes; Severe Obesity; Metabolic Surgery; Continuous Glucose Monitoring; Glucose Variability; Post-Bariatric Hypoglycemia; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CGM group (Experimental)
  Interventions: Device: Abbot Freestyle Libre CGM
- SMBG group (No Intervention)

INTERVENTIONS:
Device: Abbot Freestyle Libre CGM — Participants assigned to the CGM group will receive the Libre 2+ systems (Abbott Diabetes Care, Alameda, CA) upon randomization. This will include comprehensive training provided by a qualified healthcare professional. The training will cover detailed instructions on sensor placement, how to download and use the associated smartphone application, and guidance on interpreting the glucose data effectively. To ensure continuous and accurate monitoring, the CGM sensor will be routinely replaced every 14 days following randomization. Additionally, in the event of sensor detachment or loss, immediate replacement will be arranged to maintain uninterrupted glucose tracking. Regular sessions are conducted to analyze glucose trends, refine management strategies, and provide additional support or education on device usage.
  Arms: CGM group

SUMMARY:
Diabetes represents a significant global health burden, with its prevalence continuously rising and causing extensive impacts on individuals, healthcare systems, and society. The International Diabetes Federation (IDF) Diabetes Atlas 2021 reported a global prevalence of 10.5%, with type 2 diabetes (T2D) comprising approximately 90% of cases. In the US, diabetes prevalence stands at 11.6%, affecting roughly 38.4 million adults, with approximately 1.2 million new diagnoses each year.

Obesity, affecting over 42% of US adults-including 9.4% with severe obesity-is recognized as the primary risk factor for diabetes. Severe obesity, present in around 30% of T2D patients, markedly elevates the risk for cardiovascular disease, non-alcoholic fatty liver disease, and other comorbidities, resulting in increased mortality rates. Addressing this burden requires coordinated strategies targeting prevention, early diagnosis, effective treatment, and patient education. However, conventional management methods, such as lifestyle modifications and pharmacotherapy, often result in transient weight loss and temporary diabetes remission, with frequent relapses.

In contrast, metabolic surgery, notably Roux-en-Y gastric bypass (RYGB) and vertical sleeve gastrectomy (VSG), has emerged as a highly effective intervention for significant weight loss and durable diabetes remission, particularly among patients with severe obesity and T2D. These procedures improve metabolic outcomes beyond weight reduction, enhancing insulin sensitivity and glycemic control. Consequently, integrating metabolic surgery into standard diabetes care guidelines and expanding patient access is crucial.

Although metabolic surgery outperforms intensive medical therapy, traditional assessment methods, such as HbA1c, have notable limitations. HbA1c measures average glucose levels without capturing short-term fluctuations, glucose variability, or hypoglycemia, limiting its utility post-surgery. Continuous glucose monitoring (CGM) offers real-time, detailed insights into glucose patterns, variability, postprandial excursions, and hypoglycemia, making it highly suitable for postoperative monitoring.

CGM provides a clearer picture of immediate and long-term metabolic changes following surgery, allowing early identification of abnormal glycemic patterns influenced by surgical alterations in gastrointestinal anatomy and diet. It enables the detection of post-bariatric hypoglycemia (PBH), a recognized complication following metabolic surgery, and improves understanding of hypoglycemia unawareness-critical for enhancing patient safety and clinical outcomes.

However, current research on CGM in metabolic surgery remains limited, primarily consisting of cross-sectional or retrospective studies with small sample sizes, lacking preoperative data, and employing short monitoring periods. Therefore, robust studies such as randomized controlled trials (RCTs) are essential to validate CGM's efficacy and inform its broader adoption in clinical practice.

DETAILED DESCRIPTION:
Diabetes is a major global health concern due to its increasing prevalence, associated complications, the burden, and places on individuals, healthcare systems, and societies at large. According to the IDF Diabetes Atlas 2021, about 10.5% of the adults worldwide had diabetes, with T2D accounting for about 90% of these cases. Diabetes poses a significant health challenge in US, with approximately 38.4 million-11.6% of the US adults-diagnosed with the condition. Each year, an estimated 1.2 million adults receive a diabetes diagnosis in the US. Obesity is listed as the most important risk factor associated with diabetes. More than 42% of US are classified as obese and 9.4% have severe obesity. About 30% of patients with T2D have severe obesity. The combination of severe obesity and T2D significantly increases the risk of CVD, non-alcoholic fatty liver disease, and other comorbidities, which contribute to higher mortality rates. To tackle this heavy burden, there's a need for coordinated efforts that encompass prevention, early diagnosis, effective treatment, and patient education. The management of T2D and obesity faces several persistent challenges, including achieving sustainable weight loss and maintaining long-term diabetes remission. While lifestyle interventions and pharmacotherapy often lead to initial improvements, weight regain remains a significant issue, undermining long-term success. Similarly, diabetes remission achieved through these methods is frequently temporary, with many patients experiencing a relapse in glycemic control over time. In this context, metabolic surgery, including procedures such as Roux-en-Y gastric bypass (RYGB) and vertical sleeve gastrectomy (VSG), has emerged as one of the most effective interventions for significant weight loss and long-term diabetes remission, particularly in individuals with severe obesity and T2D. Its metabolic benefits extend beyond weight reduction, directly improving insulin sensitivity and glycemic control. Therefore, integrating metabolic surgery into treatment guidelines and expanding access to eligible patients are critical steps toward addressing the limitations of conventional approaches. While metabolic surgery has been shown to be more effective than intensive medical management for diabetes, its outcomes are often assessed using HbA1c, which has several limitations. HbA1c reflects average blood glucose levels but fails to capture glucose variability or detect hypoglycemia effectively. Additionally, it responds slowly to interventions, making it less suitable for tracking short-term changes post-surgery. These limitations have led to growing interest in CGM as a more precise tool for assessing glucose patterns after metabolic surgery. However, available data on CGM outcomes in this context remain limited, highlighting the need for further research. CGM holds significant potential for improving the assessment and management of obese patients with T2D undergoing metabolic surgery. Unlike traditional measures such as HbA1c, CGM provides real-time, continuous data on glucose levels, offering a detailed picture of glucose variability, postprandial spikes, and hypoglycemic events. This granular insight enables better tracking of short-term metabolic changes immediately after surgery and facilitates early detection of glycemic patterns that may be influenced by the changes in GI tract and dietary patterns after surgery. In the long term, CGM can monitor sustained glycemic control and identify signs of diabetes recurrence, contributing to personalized post-surgical care plans. In addition, post-bariatric hypoglycemia (PBH) is an increasingly recognized complication that can arise following metabolic and bariatric procedures. CGM will enable a better understanding of hypoglycemia unawareness, where patients fail to perceive symptoms despite critically low glucose levels. CGM may have the potential to revolutionize the management of PBH. Despite its promise, research on CGM among patients receiving metabolic surgery remains limited. Several studies have demonstrated the advantages of CGM in identifying post-bariatric hypoglycemia (Table 1). However, limitations of prior studies include their cross-sectional or retrospective design, small sample sizes, a lack of pre-surgery CGM data, and a short GDM monitoring period (most <10 days) with only one GDM measurement taken after surgery. As a result, there is a growing need for more robust studies, such as RCTs, to validate the effectiveness of this approach and optimize its integration into clinical practice.

Therefore, the investigators aim to, Aim 1: To identify the glycemic patterns by using CGM in severely obese patients with T2D receiving bariatric surgeries before and after the procedures. Hypothesis: CGM will reveal distinct glycemic patterns in obese patients with T2D undergoing metabolic surgery, with significant improvements in mean glucose control but not glycemic variability compared to baseline measures.

Aim 2: To investigate if the metrics that are derived from CGM data before and after the surgery can predict post bariatric hypoglycemia. Hypothesis: Metrics derived from CGM data, such as time in range, glycemic variability, and mean glucose levels, can reliably predict the likelihood of post bariatric hypoglycemia, with specific thresholds or patterns serving as robust predictors of long-term glycemic control.

Aim 3: To investigate the effect of CGM use on the prevention of post bariatric hypoglycemia, as well as the influence of dietary content, formulation, and patterns on glycemic responses. Hypothesis: Dietary content, formulation, and patterns significantly influence glycemic responses in obese patients with T2D, with higher fiber and protein intake, balanced macronutrient formulation, and consistent meal patterns associated with improved glycemic control and reduced risk of post bariatric hypoglycemia as measured by CGM after the surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. age 20 to 60 years
2. T2D not well controlled with medications (HbA1c >7.0%)
3. body mass index (BMI) ≥35 kg/m2
4. diabetes duration ≤ 10 years

Exclusion Criteria:

1. age <20 or ≥60 years
2. confirmed type 1 diabetes
3. pregnancy or breastfeeding
4. history of hypersensitivity to any of the components of the subcutaneous infusions
5. without access at home to a telephone or other factor likely to interfere with ability to participate reliably in the study
6. history of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer
7. patients on insulin therapy before surgery
8. patients receiving revisional surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in coefficient of variance (CV) evaluated by CGM | 9 months
  Differences in coefficient of variance (CV) evaluated by CGM

SECONDARY OUTCOMES:
Differences in HbA1c | 9 months
Total number of hypoglycemia events | 9 months
Remission rate of diabetes | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD to be shared:
  The following individual participant data will be shared upon reasonable request and approval:
  Demographic Information: Age, sex, race/ethnicity, BMI.
  Clinical Data: Baseline and follow-up clinical parameters, including diabetes diagnosis, diabetes duration, HbA1c levels, blood glucose measures, medication use, and relevant comorbidities.
  Surgical Information: Type of metabolic surgery performed, date of surgery, and perioperative outcomes.
  Continuous Glucose Monitoring (CGM) Data: Raw and analyzed CGM data including glucose variability, time in range, episodes of hypoglycemia, and hyperglycemia.
  Outcomes Data: Weight loss, diabetes remission status, insulin sensitivity measures, and occurrence of post-bariatric hypoglycemia (PBH).
  Safety Data: Adverse events related to metabolic surgery or CGM device use
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available following the publication of the primary study results. Data will be available for up to 5 years post-publication.
Access Criteria: Access to IPD requires a formal, scientifically valid request detailing the intended analyses and ethical justification. Requests will be reviewed by the original research team to ensure compliance with ethical standards and data protection regulations.

REFERENCES:
- [Background] Hanipah ZN, Schauer PR. Bariatric Surgery as a Long-Term Treatment for Type 2 Diabetes/Metabolic Syndrome. Annu Rev Med. 2020 Jan 27;71:1-15. doi: 10.1146/annurev-med-053117-123246. PMID 31986081
- [Background] Battelino T, Alexander CM, Amiel SA, Arreaza-Rubin G, Beck RW, Bergenstal RM, Buckingham BA, Carroll J, Ceriello A, Chow E, Choudhary P, Close K, Danne T, Dutta S, Gabbay R, Garg S, Heverly J, Hirsch IB, Kader T, Kenney J, Kovatchev B, Laffel L, Maahs D, Mathieu C, Mauricio D, Nimri R, Nishimura R, Scharf M, Del Prato S, Renard E, Rosenstock J, Saboo B, Ueki K, Umpierrez GE, Weinzimer SA, Phillip M. Continuous glucose monitoring and metrics for clinical trials: an international consensus statement. Lancet Diabetes Endocrinol. 2023 Jan;11(1):42-57. doi: 10.1016/S2213-8587(22)00319-9. Epub 2022 Dec 6. PMID 36493795
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] GBD 2021 US Burden of Disease and Forecasting Collaborators. Burden of disease scenarios by state in the USA, 2022-50: a forecasting analysis for the Global Burden of Disease Study 2021. Lancet. 2024 Dec 7;404(10469):2341-2370. doi: 10.1016/S0140-6736(24)02246-3. PMID 39645377

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT07095972/Prot_SAP_000.pdf